CLINICAL TRIAL: NCT06548529
Title: Al18F-HER2-BCH PET/CT to Predict Response in Bladder Cancer Patients Treated With HER2 ADC
Brief Title: HER2 Expression of HER2 Affibody-based PET/CT to Predict Response in Bladder Cancer Patients Treated With ADC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019KT114
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-06

CONDITIONS: HER2 Positive or Suspicious Positive Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Al18F-HER2-BCH PET/CT in bladder cancer patients (Experimental)
  Interventions: Radiation: HER2 expression of PET imaging

INTERVENTIONS:
Radiation: HER2 expression of PET imaging — Evaluate the diagnostic potential of HER2 imaging using 18F-labelled HER2 affibody , evaluate the predictive and prognostic value of HER2 PET imaging in bladder cancer patients treated with ADC

SUMMARY:
To use the molecular PET radionuclide (F-18) labelled HER2 Affibody to evaluate the predictive and prognostic value of HER2 expression in bladder cancer patients treated with HER2 ADC

ELIGIBILITY:
Inclusion Criteria:

1. Aged # 18 years old; ECOG 0 or 1;
2. Is unresectable or metastatic;
3. Patients with HER2 positive or suspicious positive tumors;
4. was previously treated with trastuzumab and taxane in the advanced setting or progressed within 6 months after neoadjuvant or adjuvant treatment involving a regimen including trastuzumab and taxane;
5. Has adequate cardiac, bone marrow, renal, hepatic and blood clotting functions;
6. Receives anti-HER2 ADC treatment
7. Life expectancy > 3 months

Exclusion Criteria:

1. Significant hepatic or renal dysfunction;
2. Is pregnant or ready to pregnant;
3. Cannot keep their states for half an hour;
4. Refused to join the clinical research;
5. Suffering from claustrophobia or other mental disorders;
6. Any other situation that researchers considered it unsuitable to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
SUV | 4 years
  The uptake of the tracer in the primary and metastatic tumor lesions by measuring standardized uptake value (SUV) on PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- uEXPLORER total-body PET/CT scanner (United Imaging, China), Beijing, China